CLINICAL TRIAL: NCT04398329
Title: A Phase 1b/2, Randomized, Blinded, Active-Controlled Study of Escalating Doses of HTX-034 for Postoperative Analgesia in Subjects Undergoing Unilateral, First Metatarsal Bunionectomy With Osteotomy and Internal Fixation
Brief Title: Dose-Escalation Study of HTX-034 Following Bunionectomy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HTX-034-101
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Bunions
Keywords: Analgesia; Bunionectomy
MeSH Terms: conditions — Bunion; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (5):
- Phase 1b (Cohort 1) (Experimental): Fixed dose of HTX-034.
  Interventions: Drug: HTX-034; Device: Luer lock applicator
- Phase 1b (Cohort 2) (Experimental): Individualized dose of HTX-034.
  Interventions: Drug: HTX-034; Device: Luer lock applicator
- Phase 2 (Expansion): Low Dose (Experimental): Fixed dose of HTX-034.
  Interventions: Drug: HTX-034; Device: Luer lock applicator
- Phase 2 (Expansion): High Dose (Experimental): Individualized dose of HTX-034.
  Interventions: Drug: HTX-034; Device: Luer lock applicator
- Phase 1b and Phase 2 (Active Comparator): Bupivacaine HCl.
  Interventions: Drug: Bupivacaine HCl

INTERVENTIONS:
Drug: HTX-034 — HTX-034, low dose
  Arms: Phase 1b (Cohort 1); Phase 2 (Expansion): Low Dose
Drug: HTX-034 — HTX-034, high dose
  Arms: Phase 1b (Cohort 2); Phase 2 (Expansion): High Dose
Device: Luer lock applicator — Applicator for instillation
  Arms: Phase 1b (Cohort 1); Phase 1b (Cohort 2); Phase 2 (Expansion): High Dose; Phase 2 (Expansion): Low Dose
Drug: Bupivacaine HCl — Bupivacaine HCl, 50 mg
  Arms: Phase 1b and Phase 2

SUMMARY:
This is a Phase 1b/2, randomized, blinded, active-controlled study. Phase 1b will evaluate escalating doses of HTX-034 compared with bupivacaine HCl. Phase 2 will be a dose-expansion phase to evaluate additional subjects treated with the HTX-034 dose selected based on Phase 1b compared with bupivacaine HCl.

ELIGIBILITY:
Inclusion Criteria:

* Is medically fit to undergo an elective unilateral, first metatarsal bunionectomy with osteotomy and internal fixation under regional anesthesia; no neuraxial technique (eg, no spinal, epidural, or general anesthesia).
* Has an American Society of Anesthesiologists (ASA) Physical Status of I, II, or III.
* Female subjects are eligible only if not pregnant, not lactating, not planning to become pregnant during the study; sterile, or using acceptable contraceptives.

Exclusion Criteria:

* Had contralateral foot bunionectomy in the past 3 months.
* Has a planned concurrent surgical procedure.
* Has a contraindication or a known or suspected history of hypersensitivity or clinically significant idiosyncratic reaction to required study medications.
* Has a pre-existing concurrent acute or chronic painful physical/restrictive condition expected to require analgesic treatment in the postoperative period for pain.
* Has received or is taking a contraindicated or prohibited medications.
* Received an investigational product or device in a clinical trial within 30 days or within 5 elimination half lives.
* Has a known or suspected history of drug abuse, a positive drug screen on the day of surgery, or a recent history of alcohol abuse.
* Has a history of clinically significant cardiac abnormality such as myocardial infarction within 6 months.
* Has a history of coronary artery bypass graft surgery within 12 months.
* Has a history of known or suspected coagulopathy.
* As per subject history and/or medical records, has active infection or is currently undergoing treatment for Hepatitis B, Hepatitis C, or human immunodeficiency virus (HIV).
* Has uncontrolled anxiety, psychiatric, or neurological disorder.
* Had a malignancy in the last year, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
* Has undergone 3 or more surgeries within 12 months.
* Has a known history of glucose-6-phosphate dehydrogenase deficiency.
* Has any of the following laboratory abnormalities during Screening (1 retest permitted):

  * Severe liver function impairment.
  * Severe kidney function impairment.
  * Platelet count <100,000/μL, hemoglobin <12 g/dL, or hematocrit <35%.
* Has a body mass index (BMI) >39 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent adverse events (TEAE's) (Phase 1B) | 42 days
Mean area under the curve (AUC) of the NRS scores through 72 hours (AUC0-72) for the pooled Phase 1b and Phase 2 | 7 days

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of HTX-034 | 29 days
Time of maximum plasma concentration (Tmax) of HTX-034 | 29 days
Area under the concentration-time curve from Time 0 to the time of the last quantitative concentration (AUClast) of HTX-034 | 29 days
Area under the concentration-time curve from Time 0 extrapolated to infinity (AUCinf) of HTX-034 (Phase 1B) | 22 days
Apparent terminal half-life (t½) of HTX-034 (Phase 1B) | 22 days
Mean AUC of the NRS pain intensity scores | 7 days
Total postoperative opioid consumption (in IV Morphine Milligram Equivalents) | 7 days
Proportion of subjects who are opioid-free | 14 days
Incidence of serious adverse Events (SAE's) | 42 days

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Arizona Research Center, Phoenix, Arizona
  - First Surgical Hospital, Bellaire, Texas
  - Endeavor Clinical Trials, LLC, San Antonio, Texas
  - JBR Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided